CLINICAL TRIAL: NCT03937453
Title: A PAncreatic Cancer Screening Study in Individuals With New-Onset or DeteriOrating Diabetes MEllitus (PANDOME Study)
Brief Title: A Pancreatic Cancer Screening Study in Individuals With New-Onset or Deteriorating Diabetes Mellitus
Acronym: PANDOME
Status: Recruiting | Type: Observational
Sponsor: Nuvance Health (Other)
Responsible Party: Principal Investigator, Richard Frank, Director of Cancer Research, Nuvance Health
Other Study IDs: 18-01
Record Dates: First submitted 2019-04-05; First posted 2019-05-03 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasms
Keywords: Pancreas; Cancer; Diabetes Mellitus; MRI; Early Detection
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New-Onset Diabetes Mellitus: Diabetes Mellitus diagnosed within the past 12 months
  Interventions: Diagnostic Test: MRI/MRCP
- Deteriorating Diabetes Mellitus: History of Diabetes Mellitus with recent deteriorating within the past 6 months confirmed with repeat testing and not associated with weight gain or diabetes medication non-compliance
  Interventions: Diagnostic Test: MRI/MRCP

INTERVENTIONS:
Diagnostic Test: MRI/MRCP — An MRI/MRCP with IV gadolinium contrast with high resolution imaging of the pancreas will be performed at baseline. Further imaging upon recommendation by study committee

SUMMARY:
The main goal of this study is to explore the relationship between new-onset diabetes mellitus/deteriorating diabetes and a subsequent diagnosis of pancreatic cancer. Magnetic Resonance Imaging and Magnetic cholangiopancreatography (MRI/MRCP) will be utilized to screen for early stage pancreatic cancer or precursor lesions. Participants will be asked to donate a blood sample at specific intervals for the creation of a bio-bank necessary for the development of a blood based screening test for pancreatic cancer.

DETAILED DESCRIPTION:
Individuals over 50 years of age who have developed new-onset diabetes mellitus (diagnosed within the past 12 months) or deteriorating diabetes will be recruited through the offices of primary care physicians and endocrinologists. Those meeting initial criteria will meet with a research APRN and will undergo a secondary screen to determine eligibility. Individuals enrolled in the study will undergo a five-minute psychological survey and donation of a blood sample for bio-bank analysis every 6 months for 3 years. MRI will be performed at baseline. Any abnormalities on MRI will be reviewed by a multi-disciplinary tumor board and discussed with the participant. Additional MRI will be performed on case-by-case basis

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 50 years.
* DM of Confirmed Duration: DM diagnosed within the past 12 months AND documentation of prior normal FPG, OGTT or HbA1c levels within the past 2 years. Requirement for HbA1c ≥ 6.5% OR
* DM of Unconfirmed Duration: DM diagnosed within the past 12 months BUT no prior record of normal FPG, HbA1c or OGTT within the past 2 years. Requirement for HbA1c ≥ 7.0% OR
* Transition from pre-Diabetes to Diabetes Mellitus within the past 12 months characterized by a change in the HbA1c of ≥ 0.5% OR
* DM With Only One FDR: DM diagnosed within the past 12 months that is of Confirmed or Unconfirmed Duration, in an individual with 1 FDR. Requirement for HbA1c ≥ 6.5%. OR
* Deteriorating Diabetes: DM with >2% spike in HbA1c within past 6 months confirmed with repeat testing and NOT associated with weight gain and diabetes medication non-compliance
* ECOG Performance Status of 0-1.
* No known contraindications to MRI examination or gadolinium contrast.
* Willing to undergo MRI and screening for metal implants or metal injury.
* Recent BUN and Cr
* Estimated GFR (eGFR) must be greater than 30 mL/min.
* Ability to provide informed consent.
* Willing to return to study site for all study assessments.

Exclusion Criteria:

* Prior history of pancreatic cancer.
* Presence of metastatic cancer or cancer requiring adjuvant chemotherapy within the past 5 years.
* Received chemotherapy within the past 6 months. (Hormonal therapy is allowable if the disease free interval is at least 5 years).
* Hereditary pancreatitis.
* eGFR < 30 mL/min.
* Contraindication to MRI examination or gadolinium contrast.
* Pregnant or nursing women.
* Co-morbid illnesses or other concurrent disease which, in the judgment of the clinicians obtaining informed consent, would make the participant inappropriate for entry into this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50+ years of age. New-onset diabetes mellitus (diagnosed with within the preceding 12 months) or Deteriorating diabetes mellitus (spike in HbA1c within past 6 months without weight gain and medication non-compliance)
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2028-01-19 (Estimated); Study Completion 2028-01-19 (Estimated)

PRIMARY OUTCOMES:
Early Stage Pancreatic Cancer or Precursor Lesions | Through study completion, up to 3 years
  Determine incidence of pancreatic cancer or precursor lesions in individuals with new-onset diabetes mellitus or deteriorating diabetes

SECONDARY OUTCOMES:
Relative Risk of Pancreatic Cancer Among Individuals with New-Onset Diabetes | Through study completion, up to 3 years
  Assess utility of MRI as a screening tool for pancreatic cancer and ascertain relative risk of pancreatic cancer in study population of individuals with new-onset diabetes compared to a normal population of the same age
Relative Risk of Pancreatic Cancer Among Individuals with Detiorating diabetes | Through study completion, up to 3 years
  Assess utility of MRI as a screening tool for pancreatic cancer and ascertain relative risk of pancreatic cancer in study population of individuals with deteriorating diabetes compared to a normal population of the same age

CONTACTS AND LOCATIONS:
Overall Officials: Richard Frank, MD, Principal Investigator — Nuvance Health
Locations (1):
- Nuvance Health, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed on an individual basis post submission. Requestors may be required to sign a data access agreement

REFERENCES:
- See also: More information regarding the Pancreatic Cancer Screening Study may be found here — https://www.nuvancehealth.org/about-us/research-and-innovation/cancer-research/pancreatic-cancer-research/pancreatic-cancer-screening-study